CLINICAL TRIAL: NCT01805206
Title: An Assessment of Urinary Intestinal Fatty Acid Binding Protein as a Early Predictor of Necrotizing Enterocolitis
Brief Title: Prediction of NEC With Urinary iFABP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution prior to receiving funding
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 215610
Record Dates: First submitted 2013-03-04; First posted 2013-03-06 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Prematurity; Necrotizing Enterocolitis
Keywords: Prematurity; Necrotizing Enterocolitis; Biomarkers; Intestinal Fatty Acid Binding Protein; Feeding
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- iFABP Monitored (Experimental): Subjects monitored for urinary iFABP content during the first 4-12 days of life. Enteral feedings administered when iFABP levels are normal during the first four days of life or, if elevated during the first four days of life, have normalized for five days.
  Interventions: Other: Assessment of urinary iFABP; Other: Administration of enteral feedings

INTERVENTIONS:
Other: Assessment of urinary iFABP
Other: Administration of enteral feedings

SUMMARY:
During the first four days of life, intestinal fatty acid binding protein (iFABP) is elevated in the urine of premature babies who go on to develop necrotizing enterocolitis (NEC) days to weeks later. This study aims to determine whether the withholding of feedings in babies with an elevated urinary iFABP can reduce the incidence of NEC.

DETAILED DESCRIPTION:
Necrotizing enterocolits (NEC) occurs with an incidence of 3-7% in very low birth weight (<1500g) infants and is associated with significant morbidity and mortality. Earlier detection of a subclinical prodrome in NEC might allow for the institution of measures that could prevent or attenuate the severity of disease. We have demonstrated that levels of urinary intestinal fatty acid binding protein (iFABPu), a sensitive and specific marker for intestinal mucosal injury, were elevated in the first 4 days of life in all infants who subsequently developed NEC. We hypothesize that, in the context of an elevated iFABPu in the neonatal period, a significant proportion of NEC cases could be averted by not initiating feedings.

The proposed study will be a three-year prospective trial of iFABPu monitoring during the neonatal period in 220 infants of gestational age less than 33 weeks. Urine will be collected in 12-hour aliquots over the first four days of life and the iFABPu will be measured. On the afternoon of day of life four, infants in whom iFABPu exceeded 1000 pg/ml at any time will be continued with no feedings, iFABPu will continue to be measured, and trophic, breast milk feedings will only be initiated after iFABPu has normalized for five days. Infants with non-elevated iFABPu over the first four days of life will have feedings initiated on day of life four, in the absence of other contraindications. All subjects will have urine collected daily over their entire hospital stay for iFABPu assay. However, after the active study period (after feedings have been initiated) iFABPu findings will not be communicated to the physicians caring for the subjects, but will be evaluated retrospectively in order to better define the utility of iFABPu as a marker for impending NEC later in newborn life.

If iFABPu monitoring is shown to be effective in reducing the incidence of NEC it would revolutionize the care of premature infants by providing physicians with a tool that would permit feeding decisions to be based directly upon the viability of the intestine, rather than intuition.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age less than 33 weeks
* Admission to Loma Linda University Children's Hospital NICU within 48 hours of life

Exclusion Criteria:

* Anuria
* Congenital gastrointestinal anomaly

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of necrotizing enterocolitis | 90 days

SECONDARY OUTCOMES:
Time to caloric goal for enteral feedings | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gollin, MD, Principal Investigator — Loma Linda University School of Medicine
Locations (1):
- Loma Linda University Children's Hospital, Loma Linda, California, United States

REFERENCES:
- [Background] Mannoia K, Boskovic DS, Slater L, Plank MS, Angeles DM, Gollin G. Necrotizing enterocolitis is associated with neonatal intestinal injury. J Pediatr Surg. 2011 Jan;46(1):81-5. doi: 10.1016/j.jpedsurg.2010.09.069. PMID 21238645
- [Background] Stadie D, Boskovic DS, Plank MS, et al. Elevated urinary intestinal fatty acid binding protein precedes clinical indicators of necrotizing enterocolitis. JSR 179:319, 2013.